CLINICAL TRIAL: NCT01107236
Title: A Phase 2, Single-center, Randomized, Double-blind, Placebo- and Active-controlled, Parallel-group Study of a Single Dose of IW-6118, in Patients Undergoing Third Molar Extraction
Brief Title: Study to Evaluate Efficacy and Safety of IW-6118 in Patients Undergoing Third Molar Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-109-201
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Healthy subjects
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- IW-6118 (Experimental)
  Interventions: Drug: IW-6118
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo
- Naproxen Sodium (Active Comparator)
  Interventions: Drug: Naproxen Sodium

INTERVENTIONS:
Drug: IW-6118 — Single dose
  Arms: IW-6118
Drug: Matching Placebo — Single dose of matching placebo for IW-6118 and/or matching placebo for naproxen sodium
  Arms: Placebo
Drug: Naproxen Sodium — Single dose
  Arms: Naproxen Sodium

SUMMARY:
The purpose of this study is to assess the safety of IW-6118 when administered as a single oral dose to patients undergoing third molar extraction. Efficacy will be assessed in an exploratory manner.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 30 years old at time of screening;
* BMI > 18.5 and < 30.0;
* In overall good health with no clinically-significant laboratory, ECG, or physical exam findings;
* Patient requires two ipsilateral third molar extractions of which one must be a full or partial bony mandibular impaction;
* Women of childbearing potential must have a negative pregnancy test and must agree to use double-barrier contraception;
* Other inclusion criteria per protocol.

Exclusion Criteria:

* History of any clinically-significant medical condition;
* Previous usage of prescription, OTC, or investigational drugs as per protocol requirements;
* Inadequate levels of pain to be included in the study;
* Other exclusion criteria per protocol.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety Assessments | Duration of the Study
  Adverse events, vital signs, laboratory parameters, and ECGs will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Ironwood Investigational Site, Salt Lake City, Utah, United States